CLINICAL TRIAL: NCT01010594
Title: Two Pieces of Fruit to Type 2 Diabetics?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI changed job and project was not economically viable and therefor terminated
Sponsor: Hospitalsenheden Vest (Other)
Responsible Party: Principal Investigator, Allan Stubbe Christensen, MHSc, RD, Hospitalsenheden Vest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-20090183
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fruit restricted (Active Comparator): Type 2 diabetics are advised to restrict their fruit intake to two pieces or less daily.
  Interventions: Behavioral: dietary treatment
- Fruit ad libitum (Active Comparator): Type 2 diabetics are advised to eat at least two pieces of fruits daily
  Interventions: Behavioral: dietary treatment

INTERVENTIONS:
Behavioral: dietary treatment — A standard dietary treatment except that they are advised to restrict their fruit intake.
  Arms: Fruit restricted
Behavioral: dietary treatment — A standard dietary treatment.
  Arms: Fruit ad libitum

SUMMARY:
It has been questioned whether patients with type 2 diabetes who are advised to restrict their fruit consumption to two or less pieces of fruits daily have better outcomes (HbA1c, body weight, fruit intake and serum lipids) after three months compared to patients with type 2 diabetes who are advised to eat at least two pieces of fruits.

To the investigators' knowledge, no randomized controlled trial has evaluated this.

The investigators therefore perform a randomized controlled trial including 76 patients with type 2 diabetes to investigate this.

The investigators' hypothesis is that:

Type 2 diabetics who are advised to restrict their fruit consumption have the same Hba1c three months after an initially dietary treatment as type 2 diabetics who are advised not to restrict their fruit consumption.

ELIGIBILITY:
Inclusion Criteria:

* patients refered from a general practitioner

Exclusion Criteria:

* no Hba1c when refered
* Hba1c lower than 5% or higher than 12%
* patients that require a translator
* patients with severe cardiovascular, renal or endocrine disease
* psychiatric patients
* pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in Hba1c | three months

SECONDARY OUTCOMES:
change in bodyweight | three months
change in serum lipids | three months
change in fruit intake | three months

CONTACTS AND LOCATIONS:
Overall Officials: Allan S Christensen, MHSc, Principal Investigator — The Department of Endocrinology and Metabolism, Aarhus University Hospital
Locations (1):
- Department of nutrition, Regional Hospital West Jutland, Holstebro, Holstebro, Denmark

REFERENCES:
- [Result] Christensen AS, Viggers L, Hasselstrom K, Gregersen S. Effect of fruit restriction on glycemic control in patients with type 2 diabetes--a randomized trial. Nutr J. 2013 Mar 5;12:29. doi: 10.1186/1475-2891-12-29. PMID 23497350